CLINICAL TRIAL: NCT06260020
Title: Development and Validation of a Comprehensive Module for Management of Sleep Disorders in Children With Autism Spectrum Disorder Aged 4-10 Years: a Pre and Post Intervention Study
Brief Title: Development and Validation of a Comprehensive Module for Management of Sleep Disorders in ASD Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Professor, All India Institute of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IECPG-463/24.08.2023
Record Dates: First submitted 2024-01-18; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Sleep Disorder; Autism Spectrum Disorder; Polysomnography; Actigraphy; Children; Behavior Therapy
Keywords: ASD; PSG; CSHQ; Actigraphy; sleep
MeSH Terms: conditions — Sleep Wake Disorders; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Pre and post intervention study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children [4-10 years] with ASD with sleep disorder (Experimental): Development of module by Delphi method:components of Module include Behavioural intervention Modifying stimulus by change in location,using bedtime stories. Giving schedules to activities which interfere with sleep before bedtime. Using a bedtime pass to allow child to make a prefixed number of requests for parental attention while in bed.
  Giving sleep items like cuddle toys to replace parental presence. Gradually delaying the bedtime so the child feels urge to sleep. Sleep hygiene by providing suitable environment to sleep, proper bedtime routine, sleep wake schedules Providing rewards for following good bedtime routine as positive reinforcement. Pharmacological intervention Sleep disorders due to underlying ENT, pulmonary conditions, to be treated as per standard protocol Usage of melatonin if required for sleep onset difficulty An 80%agreement over an intervention will be included in the module
  Interventions: Behavioral: Comprehensive module for management of sleep disorders[Behavioral and pharmacological therapy]

INTERVENTIONS:
Behavioral: Comprehensive module for management of sleep disorders[Behavioral and pharmacological therapy] — Development of module by Delphi method:components of Module include Behavioural intervention Modifying stimulus by change in location,using bedtime stories. Giving schedules to activities which interfere with sleep before bedtime. Using a bedtime pass to allow child to make a prefixed number of requests for parental attention while in bed.
  Giving sleep items like cuddle toys to replace parental presence. Gradually delaying the bedtime so the child feels urge to sleep. Sleep hygiene by providing suitable environment to sleep, proper bedtime routine, sleep wake schedules Providing rewards for following good bedtime routine as positive reinforcement. Pharmacological intervention Sleep disorders due to underlying ENT, pulmonary conditions, to be treated as per standard protocol Usage of melatonin if required for sleep onset difficulty An 80%agreement over an intervention will be included in the module

SUMMARY:
Sleep disorder in autism children is common and it affects the physical, behavior and mental health. There is lack of comprehensive management program/module to treat the sleep disorders in children with ASD. Limited studies evaluating the utility of actigraphy to diagnose sleep disorders in ASD and its validation with PSG are present. Rationale of this study is to develop the comprehensive module and validate it for children with autism spectrum disorders, so as to improve the behavioral outcomes as well. This study also helps to utilize actigraphy as a modality to diagnose sleep disorders in children with autism spectrum disorder as performing PSG in these children is cumbersome and difficult as ASD children tend to have sensory abnormalities.

DETAILED DESCRIPTION:
Development of module for management of sleep disorders in children with ASD will be done by Delphi method:

Proposed components of Module include

Behavioral intervention

1. Modifying stimulus by change in location of sleep onset, using bedtime stories.
2. Giving schedules to activities which interfere with sleep before bedtime itself so they don't disturb the sleep onset now .
3. Using a bedtime pass which allows children to make a predetermined number of requests for parental attention while in bed.
4. Giving sleep items like cuddle toys to replace the parental presence
5. Delaying the bedtime so the child feels urge to sleep and slowly decreasing that time
6. Sleep hygiene by providing suitable environment for child to sleep, providing proper bedtime routine, sleep wake schedules
7. Providing rewards for children who followed the good bedtime routine as positive reinforcement.

Pharmacological intervention

1. For children diagnosed with sleep disorders due to underlying ENT, pulmonary conditions, to treat them accordingly as per standard protocol available.
2. Usage of melatonin if required for sleep onset difficulty

An 80% agreement over an intervention will be included in the module. The module will be developed within 3 months and ethical approval will be taken for application of this intervention.

Children aged 4 to 10 years attending Pediatric autism clinic and diagnosed with ASD using DSM V criteria, who are on follow up with behavioral therapy at least for 6 months will be included in the study. On routine comprehensive evaluation those children with refractory epilepsy and ASD children with tuberous sclerosis, fragile X syndrome and Down syndrome and metabolic disorders will be excluded.

The child will undergo screening for identification of sleep disorders initially.

They will be called around 11 am on the day of assessment, from 12 noon they will be made to wear the actigraphy watch on the non-dominant wrist.

They will undergo evaluation on CSHQ, half and hour before the stipulated bedtime, PSG electrodes will be attached till lying on bed at the night time, the actigraphy parameters will be recorded as daytime data, once on the bed at night, the data will be recorded as nocturnal actigraphy data. The PSG electrodes will be removed next morning immediately after the child gets up from sleep. Actigraphy watch will be removed at 12 noon the next day.

The CSHQ will be administered by the principal investigator in Hindi or English.

Parents will be asked to answer the questions based on the sleep habits of the child based on the past week. In case the last week was unusual for a specific reason the questions were answered with respect to the most recent typical week Appointment for overnight PSG will be given as per the convenience of the family.

Parents will be advised to continue the child's usual pattern of sleep prior to the test.

For children who are on pharmacological therapy for seizures and behavioral issues, drugs will be continued so as to not interfere with the child's treatment and conform to ethics.

The parents will be told to bring the child on the day of the study with his or her night clothes along with pillows, bedsheets and any other sleep association objects that the child wanted.

The parents will be shown the laboratory once before the actual testing. This will help them in replicating the child's routine sleeping pattern as far as possible in the PSG lab on the night of testing.

Standard overnight multichannel PSG evaluation will be performed with Philips Respironics Alice 6 LDxS PSG system with Axis 5521 PTZ high-resolution camera.

PSG scoring and reporting will be done according to American Academy of Sleep Medicine Manual (version 2.5) and International Classification of Sleep Disorders -3 manual.

The PSG record will be analyzed by Pediatric neurology faculty who are blinded to clinical status and Actigraphy scoring and reporting will be done.

Complete evaluation of behavior (ATEC, CBCL, CARS-2, sensory profile, DP-3 and ABC) will be done for all children undergoing screening polysomnography, actigraphy on the same day.

CARS is done to estimate the severity of autism. It is different for high functioning children (IQ >80, age >6 years with fluent speech), with scores of 15-27.5 being minimal; 28-33.5 mild to moderate; and more than 34 is severe. For other children (age <6 years, without fluent speech) score of 15-29.5; 15-27.5(age for 13+,IQ<80) is minimal, 30-36.5 (age <6 years, without fluent speech) ;28-34.5(age for 13+,IQ<80) is mild to moderate and (age <6 years, without fluent speech) score of 37 and higher , score of 35 and higher (age for 13+,IQ<80) shows severe symptoms of Autism Spectrum Disorder. The CARS is a 15-item scale used to grade the severity of autism in 14 behavioral domains.

CBCL is used for determining the behavioral comorbidities. The CBCL assesses behavior in 11 domains and there are two sets of questionnaires, one for 1.5 to 5 years of age and another for 5 to 18 years of age which is separate for boys and girls.

Development Profile 3 (DP3) is used to estimate the development or intelligent quotient. The DP3 assesses DQ/IQ in 5 domains (Physical behavior, Adaptive Behavior, Cognition, Social Emotional and Communication) by parental reporting as well as direct observation.

The Autism Treatment Evaluation Checklist (ATEC) was designed to assist parents, physicians and researchers to evaluate virtually any treatment for autism. It includes scoring in Speech/ Language/ Communication sociability, sensory and cognitive awareness, health/physical/behavior.

The Autism Behavior Checklist (ABC) was designed to offer a method to more objectively identify autism in children. The scale utilizes an observer's rating of the child's behavior to quantify behaviors typically associated with Autism. The ABC was developed as a clinical measure to screen for autism in individuals 3-35 years of age. The scale was developed in 1980 and has not undergone revision since then. The ABC consists of 57 items and 5 scales (1) Sensory, (2) Relating, (3) Body and Object use, (4) Language and (5) Social and Self-help.

If the child is found to have sleep disorder according to ICSD -3 criteria, then they will be enrolled in the study after informed consent to undergo intervention.

They will be given module-based intervention according to the disorder child is found to have.

They will be followed up telephonically every 2 weeks and in OPD/Clinic every 4 weeks to ensure compliance with intervention.

After 6 months of intervention, CSHQ, PSG and actigraphy evaluation of behavior (ATEC, CBCL, CARS-2, sensory profile, DP-3 and ABC) will be repeated in the same method used before giving intervention.

Pre and post CSHQ scores, actigraphy and polysomnography, behavioral scores will be compared , and correlation between actigraphy and polysomnography will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 4-10 years with diagnosis of ASD and ICSD based sleep disorder
2. At-least 6 months of behavioral therapy and follow-up at AIIMS

Exclusion Criteria:

1. Refractory epilepsy
2. Secondary causes of ASD like Fragile-X Syndrome, Down Syndrome, Tuberous sclerosis
3. ASD with metabolic disorders

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Development of comprehensive module for management of sleep disorders in autism spectrum disorders | 3 months from onset of study
  The comprehensive module will be developed for management of sleep disorders. The proposed components in the module are Behavioral intervention like modifying stimulus by change in location of sleep onset,Giving schedule activities which interfere with sleep before bedtime,Using a bedtime pass which allows children to make a predetermined number of requests for parental attention while in bed,Giving sleep items,Delaying the bedtime,Sleep hygiene by providing suitable environment for child to sleep, providing proper bedtime routine , sleep wake schedules,Providing rewards as positive reinforcement.Pharmacological intervention to treat them accordingly as per standard protocol available,The components of the module will be decided based on Delphi method. Experts opinion will be taken and comprehensive module will be developed accordingly.
To validate the above module in children of ASD with sleep disorders by measuring change in Children's Sleep Habits Questionnaire(CSHQ) score pre and post intervention. | From baseline to 6 months
  The CSHQ is a parent-rated questionnaire comprised of 45 items; 33 scored questions, and 7 additional items intended to provide other relevant information pertaining to sleep behavior (e.g., nocturnal body pains) Each scored question is rated on a 3-point scale as occurring "usually" (i.e., 5-7 times within the past week), "sometimes" (i.e., 2-4 times within the past week), or "rarely" (i.e., never or 1 time within the past week).
  A number of items on the questionnaire are reverse-scored, so that higher scores consistently indicate problem behaviors.
  Ratings are combined to form eight subscales: Bedtime Resistance, Sleep Onset Delay, Sleep Duration, Sleep Anxiety, Night Wakings, Parasomnias, Sleep Disordered Breathing, and Daytime Sleepiness.
  A Total Sleep Disturbances score is calculated as the sum of all CSHQ scored questions, and can range from 33 to 99.
To validate the above module in children of ASD with sleep disorders by comparing sleep efficiency | From baseline to 6 months
  Change in sleep efficiency (%) as measured by PSG and actigraphy pre and post intervention.
To validate the above module in children of ASD with sleep disorders by comparing change in sleep onset latency | From baseline to 6 months
  Change in sleep onset latency(time duration)as measured by PSG and actigraphy pre and post intervention.

SECONDARY OUTCOMES:
To evaluate the agreement of actigraphy with polysomnography in sleep efficiency for evaluation of sleep disorders in children with autism spectrum disorder | 6 months
  Agreement between PSG and actigraphy in sleep efficiency (%) using Intraclass Correlation Coefficient and Lin's Concordance Correlation Coefficient Agreement between PSG and actigraphy in sleep efficiency (%) and sleep onset latency(duration) using Intraclass Correlation Coefficient and Lin's Concordance Correlation Coefficient
Change in autism severity using ATEC (Autism treatment evaluation checklist) score | 6 months
  Change in scores of ATEC (Autism treatment evaluation checklist) pre and post intervention ATEC is comprised of four subscales: (1) Speech/Language/Communication, (2) Sociability, (3) Sensory/Cognitive Awareness, and (4) Health/Physical/Behavior. These four subscales are used to calculate a total score that ranges from 0 to 179. A lower score indicates less severe symptoms of (Autism Spectrum Disorder)ASD and a higher score correlates with more severe symptoms of ASD.
To evaluate the agreement of actigraphy with polysomnography in determining sleep onset latency duration for evaluation of sleep disorders in children with autism spectrum disorder | 6 months
  Agreement between PSG and actigraphy in sleep onset latency (duration )using Intraclass Correlation Coefficient and Lin's Concordance Correlation Coefficient
Change in autism severity using CBCL (child behavior checklist) behavioral scales. | 6 months
  Change in scores of CBCL (child behavior checklist) pre and post intervention. CBCL is used for determining the behavioral comorbidities. The CBCL assesses behavior in 11 domains and there are two sets of questionnaires, one for 1.5 to 5 years of age and another for 6 to 18 years of age which is separate for boys and girls.The T- score of less than 65 is normal,65-70 is borderline t score, more than 70 is clinical range.
Change in autism severity using CARS-2(childhood autism rating scale -2). | 6 months
  Change in CARS-2(childhood autism rating scale -2) score pre and post intervention.
  CARS is done to estimate the severity of autism. It is different for high functioning children (IQ >80, age >6 years with fluent speech) , with scores of 15-27.5 being minimal ; 28-33.5 mild to moderate; and more than 34 is severe. For other children (age <6 years, without fluent speech) score of 15-29.5; 15-27.5(age for 13+,IQ<80) is minimal, 30-36.5 (age <6 years, without fluent speech) ;28-34.5(age for 13+,IQ<80) is mild to moderate and and (age <6 years, without fluent speech) score of 37 and higher , score of 35 and higher (age for 13+,IQ<80) shows severe symptoms of Autism Spectrum Disorder.The CARS is a 15-item scale used to grade the severity of autism in 14 behavioral domains.
Change in autism severity using Development Profile 3 (DP3) | 6 months
  Change in Development Profile 3 (DP3) score pre and post intervention. The DP3 assesses DQ/IQ in 5 domains (Physical behavior, Adaptive Behavior, Cognition, Social Emotional and Communication) by parental reporting as well as direct observation.
Change in autism severity using sensory profile. | 6 months
  Change in sensory profile score pre and post intervention. Sensory profile include Tactile (touch),Gustatory (taste),Olfactory (smell),Visual (sight),Auditory (hearing),Proprioceptive (body awareness),Vestibular (movement/balance).Child will be assesed in the above mentioned components and score will be given accordingly. Maximum score of 190 is given.
Change in autism severity using Autism Behaviour Checklist (ABC) score | 6 months
  Change in Autism Behaviour Checklist (ABC) score pre and post intervention. The ABC is a 57-item behavior rating scale assessing the behaviors and symptoms of autism for children 3 and older. The instrument consists of a list of 57 questions divided into five categories: (1) sensory, (2) relating, (3) body and object use, (4) language, and (5) social and self-help. Each item has a weighted score ranging from 1 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Sheffali Gulati, MD, Principal Investigator — All India Institute of Medical Sciences

IPD SHARING:
Plan to Share IPD: No